CLINICAL TRIAL: NCT00443274
Title: Breast Implant Follow-up Study: A Long-term Observational Study of the Safety of Allergan Silicone Gel-filled Breast Implants as Compared Both to Saline-filled Breast Implants and to National Norms (410-arm)
Brief Title: Safety Follow-up Study in Subjects With Silicone Gel-filled Breast Implants as Compared Both to Saline-filled Breast Implants and to National Norms
Acronym: BIFS
Status: Active, not recruiting | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: BIFS001; CMO-EPI-PLS-0536 (Other: AbbVie)
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Other: NBIR - US National Breast Implant Registry — NBIR is intended to be a surveillance tool to track patient safety and real-world outcomes associated with breast implants used for aesthetic or reconstructive purposes..
Device: 410 Arm — Anatomically shaped silicone gel-filled breast implants.
Device: BIFs - Breast Implant Follow-Up Study — Round silicone gel-filled breast implants and saline-filled breast implants

SUMMARY:
Ten year safety study examining rates of rare adverse events, child bearing issues, effects of mammography, MRI compliance and results, and long-term benefit of silicone-filled breast implants.

ELIGIBILITY:
Inclusion Criteria:

Screening Criteria

1. Female

   1. age 18 years or older who is a candidate for breast reconstruction (primary or revision) with Allergan silicone implants or saline breast implants (controls) OR
   2. age 22 or older who is a candidate for breast augmentation (primary or revision) with Allergan silicone implants or saline breast implants (controls)
2. Exhibit fluency and literacy in English or Spanish

Enrollment Criteria

1. Have satisfied all the inclusion and none of the exclusion criteria
2. Have completed the implant surgery
3. Have only one breast implant or have matching breast implants (i.e., both Round Responsive, both Style 410, or both saline) following their qualifying surgery. In the case of silicone, the device(s) must be manufactured by Allergan.
4. Are free of all target diseases at baseline (410 arm only)
5. Have signed the informed consent form, documenting agreement to participate in all required follow-up interviews by internet, phone, or mail and authorizing health care providers to release medical records to study personnel, and have completed the baseline questionnaire prior to implant surgery (prospectively enrolled subjects)

For retrospectively enrolled subjects into the 410 arm, in addition to the above, these criteria also apply:

1. Received 1 or 2 Style 410 implants between 2015 and 2019
2. Willing to complete baseline questionnaire at time of enrollment

Continuation Criteria (BIFS Arm Only)

1. Have completed baseline and years 1, 2, 3 and 4 follow-up questionnaires available (including the Satisfaction with Breasts and Psychosocial Well-Being modules of the BREAST-Q)
2. Met all enrollment criteria, specifically the minimum age requirements for silicone implants (18 or older for reconstruction subjects and 22 or older for augmentation subjects), and were free of all target diseases at baseline
3. Were enrolled at a site that was selected in the cluster sampling to continue in the BIFS arm

Exclusion Criteria:

1. Are transgender
2. If a saline implant subject, have a current or past unilateral or bilateral silicone gelfilled breast implant
3. Investigator decision that subject is not a suitable candidate for a long-term observational study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast implants for augmentation, reconstruction, or revision of augmentation or reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 56460 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk rates of adverse events of high clinical interest (eg, cancers, neurological diseases, connective tissue diseases) assessed by the investigator | 10 Years
Risk rates of common complications of breast surgery (eg, capsular contracture, implant rupture/deflation) assessed by the subject and investigator | 10 Years
Re-operations | 10 Years
  Rates of reoperation reported by subjects and by investigators at office visits

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (1):
- Southwest Plastic Surgery /ID# 240510, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Singh N, Picha GJ, Murphy DK. Natrelle Silicone Breast Implant Follow-Up Study: Demographics, Lifestyle, and Surgical Characteristics of More Than 50,000 Augmentation Subjects. Plast Reconstr Surg. 2016 Jan;137(1):70-81. doi: 10.1097/PRS.0000000000001851. PMID 26710009